CLINICAL TRIAL: NCT03032575
Title: SEARCH Thailand and Thai Red Cross AIDS Research Centre
Brief Title: Anal HPV Infection and Risk for Anal High-grade Squamous Intraepithelial Lesion Among Thai MSM With Acute HIV Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Collaborators: SEARCH Research Foundation (Other); amfAR, The Foundation for AIDS Research (Other); TREAT Asia (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HPV in MSM with AHI
Record Dates: First submitted 2017-01-17; First posted 2017-01-26 (Estimated); Last update posted 2024-11-25 (Actual); Status verified 2024-04

CONDITIONS: Human Papillomavirus Infection
Keywords: HIV
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sample size 100 (Other): Study Design: This is a prospective observational cohort of Thai MSM who initiated ART at the time of AHI, defined as the first 30 days after HIV acquisition (Fiebig stages 1 through 5). Volunteers will be examined at baseline to determine the prevalence of HPV infection and HSIL at HIV diagnosis. They will then be followed longitudinally for new incidence of HPV and HSIL, as well as progression or regression of existing lesions.
  Interventions: Behavioral: SEARCH010/RV254

INTERVENTIONS:
Behavioral: SEARCH010/RV254

SUMMARY:
1. To determine the prevalence and incidence of anal HSIL and associated risk factors among MSM who initiate ART during AHI.

DETAILED DESCRIPTION:
Anal human papillomavirus (HPV) infection is very common in men who have sex with men (MSM).1-3 HIV-positive MSM have a higher prevalence of anal HPV infection than HIV-negative MSM and are more likely to have infection with multiple HPV types.1,2 Spontaneous clearance of anal HPV infection is less common among HIV- positive compared with HIV-negative MSM.2 Persistent anal HPV infection, particularly with high-risk HPV types, is an important risk factor for the development of anal cancer.4-6 The incidence of anal cancer among HIV-positive MSM is very high, ranging from 75 to 137 per 100,000 person-years, and is five times higher than that in HIV-negative MSM.7-10 Anal high-grade squamous intraepithelial lesion (HSIL) is the putative precursor of anal cancer.11-13 Anal squamous intraepithelial lesion has a dynamic picture of temporal progression and regression, but HSIL is much less likely to regress than low-grade squamous intraepithelial lesion (LSIL).10,14 A recent systematic review and meta-analysis showed the pooled prevalence of anal HSIL to be 29.1% in HIV-positive MSM and 21.5% in HIV-negative MSM.15 Anal HSIL incidence ranged from 8.5 to 15.4% per year in HIV-positive MSM and 3.3 to 6.0% per year in HIV-negative MSM. Although data are limited, previous studies have shown a 9-15% progression rate from anal HSIL to anal cancer during a median follow-up of 3 - 5 years. 11-13 Previous research at the Thai Red Cross AIDS Research Centre has demonstrated high rates of HPV infection and anal HSIL among Thai MSM, with HIV-positive MSM disproportionately affected. Prevalence of anal infection with high-risk HPV types was 57.5% in HIV-positive and 36.6% in HIV-negative MSM (p = 0.008).16 Prevalence of anal HSIL was 18.9% in HIV-positive MSM and 11.4% in HIV-negative MSM (p = 0.1), while incidence of anal HSIL over 12 months was 29% and 8%, respectively (p=0.001).17 HIV-positive MSM in that study, however, were mainly naïve to antiretroviral therapy (ART) at enrollment (87% not on ART) and only 10% had undetectable HIV viral load at baseline.

It is not clear if the higher rates of HPV infection and persistence of infection are due to HIV infection or to different risk behavior among HIV-positive MSM. Data are inconclusive on whether the use of ART has an effect on anal HPV infection among HIV-positive MSM.18-19 Furthermore, there is no data on the effect that "early diagnosis" of HIV infection and "early treatment" with ART might have on incidence and persistence of HPV infection or on the development of anal HSIL.

We propose a longitudinal, observational study of HPV infection and anal HSIL among HIV-positive Thai MSM who initiate ART during acute HIV infection (AHI). The hypothesis is that early HIV diagnosis and early ART within the first 4 weeks of infection will mitigate immunological and virological factors that increase HPV persistence and anal HSIL incidence in HIV-positive MSM such that these measure will be significantly lower when compared to historical controls of chronically-infected HIV-positive Thai MSM.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or above.
2. Born biological male.
3. Self-identifies as MSM or transgender woman.
4. Enrolled in the SEARCH010/RV254 cohort.
5. In the stage of acute HIV infection diagnosed within 7 days (Fiebig I-V).
6. Agrees to start ART during acute HIV infection.
7. Had sex with a male partner at least once in the previous 3 months
8. Consents to participate in the study

Exclusion Criteria:

1. Any history of previous HSIL diagnosis or treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2023-10 (Actual)

PRIMARY OUTCOMES:
The prevalence and incidence of anal HSIL among MSM who initiate ART during AHI will be lower than among chronically-infected HIV-positive MSM, Anal HSIL is diagnosed based on histology specimen and cytology (2001 Bethesda system) | 12 months
  The prevalence of anal HSIL and the incidence of anal HSIL during the follow-up period. Anal HSIL is diagnosed based on histology specimen. A composite anal HSIL outcome (including both cytologic HSIL/ASC-H and histologic HSIL) will also be used.
  Incidence of HSIL during the follow-up period will be calculated as the number of new diagnoses per person time at risk. 95% confidence intervals (CI) will be calculated assuming a Poisson distribution. Cox proportional hazards regression will be used to identify factors associated with incident HSIL.

CONTACTS AND LOCATIONS:
Overall Officials: Nittaya Phanuphak, M.D.,Ph.D., Principal Investigator — The Thai Red Cross AIDS Research Centre
Locations (1):
- The Thai Red Cross AIDS Research Centre, Pathum Wan, Bangkok, Thailand

REFERENCES:
- [Derived] Thitipatarakorn S, Teeratakulpisarn N, Nonenoy S, Klinsukontakul A, Suriwong S, Makphol J, Hongchookiat P, Chaya-Ananchot T, Chinlaertworasiri N, Mingkwanrungruang P, Sacdalan C, Poltavee K, Pankam T, Kerr SJ, Ramautarsing R, Colby D, Phanuphak N. Prevalence and incidence of anal high-grade squamous intraepithelial lesions in a cohort of cisgender men and transgender women who have sex with men diagnosed and treated during acute HIV acquisition in Bangkok, Thailand. J Int AIDS Soc. 2024 May;27(5):e26242. doi: 10.1002/jia2.26242. PMID 38695517